CLINICAL TRIAL: NCT05206799
Title: A Multi-centre Clinical Study of Hemorrhage Rate After Coblation Tonsillectomy in Children
Brief Title: The CMCPCTH Research in Chinese Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Children's Hospital (Other)
Collaborators: Sichuan provincial maternity and child health care hospital (Unknown); Maternity and Child Health Care Hospital of Pingdingshan City (Unknown); Shanxi Provincial Maternity and Children's Hospital (Other); The Children's Hospital of Xi'an City (Unknown); Xiamen Children's Hospital (Other); Anyang Maternal and Child Health Care Center (Unknown); Ningbo Women & Children's Hospital (Other); Children's Hospital of Chongqing Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Maternity and Child Health Care Hospital of Tangshan city (Unknown); Children's Hospital Affiliated to Kunming Medical University (Unknown); Materal and Child Health Hospital of Hubei Province (Unknown); Hunan Children's Hospital (Other Government); Zhengzhou Children's Hospital, China (Other); The Children's Hospital Zhejiang University Shcool of Medicine (Unknown); Tianjin Children's Hospital (Other); Chengdu Women's and Children's Central Hospital (Other); Shenzhen Hospital of Southern Medical University (Other); Yuying Children's Hospital, second Affiliated Hospital of Wenzhou Medical University (Unknown); Jinan children's hospital (Unknown); People's Hospital of Hunan Provincial (Unknown); First People's Hospital of Foshan (Other); Jiangxi Children's Hospital (Unknown); Dalian Women and Children medical Center (Group) (Unknown); Wuxi Women's & Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021R096-E01
Record Dates: First submitted 2022-01-12; First posted 2022-01-25 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-01

CONDITIONS: Tonsillectomy; Child; Postoperative Hemorrhage
Keywords: Tonsillectomy; child; Postoperative Hemorrhage; low-temperature plasma radiofrequency ablation
MeSH Terms: conditions — Postoperative Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To obtain hemorrhage rate after coblation tonsillectomy, and to investigate risk factors of hemorrhage after coblation tonsillectomy in children.

DETAILED DESCRIPTION:
This study is a prospective and multi-centre trail in China. It intends to enroll 25000 patients underwent coblation tonsillectomy in 22 clinical centers in China. Hemorrhage rate and risk factors of hemorrhage after coblation tonsillectomy will be investigated through questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. under 18 years old;
2. Clear indications for tonsill surgery;
3. No clear contraindications for tonsill surgery;
4. Parents of the children patients accept surgical treatment;
5. Parents of the children patients able to cooperate with the visit and follow-up.

Exclusion Criteria:

1. Children patients with a history of adenoid or tonsillectomy surgery;
2. Associated with refractory bleeding diseases;
3. Combined with cleft palate;
4. Down syndrome, Prader-Willi syndrome (PWS) or other chromosomal abnormalities;
5. Neuromuscular diseases (including cerebral palsy);
6. Other diseases that affect physical health, such as severe heart disease, kidney disease, lung disease, etc;
7. Contraindications to surgery and anesthesia;
8. Unable to obtain informed consent.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Enrolled patiens are children who underwent coblation tonsillectomy from multi-centers in different provinces of China.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-01-14 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
hemorrhage rate after coblation tonsillectomy | 3 weeks after surgery
  hemorrhage rate after coblation tonsillectomy in children within 3 weeks
risk factors of hemorrhage after coblation tonsillectomy | 3 weeks after surgery
  risk factors of hemorrhage after coblation tonsillectomy in children

CONTACTS AND LOCATIONS:
Overall Officials: xiaoyan Li, PhD, Study Director — Shanghai Children's Hospital
Locations (1):
- Children's Hospital of Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yiu Y, Mahida JB, Cooper JN, Elsey NM, Deans KJ, Minneci PC, Merrill TB, Tobias JD, Elmaraghy CA. The effect of perioperative dexamethasone dosing on post-tonsillectomy hemorrhage risk. Int J Pediatr Otorhinolaryngol. 2017 Jul;98:19-24. doi: 10.1016/j.ijporl.2017.04.033. Epub 2017 Apr 24. PMID 28583496
- [Background] Sarny S, Ossimitz G, Habermann W, Stammberger H. Hemorrhage following tonsil surgery: a multicenter prospective study. Laryngoscope. 2011 Dec;121(12):2553-60. doi: 10.1002/lary.22347. PMID 22109752
- [Background] Soderman AC, Odhagen E, Ericsson E, Hemlin C, Hultcrantz E, Sunnergren O, Stalfors J. Post-tonsillectomy haemorrhage rates are related to technique for dissection and for haemostasis. An analysis of 15734 patients in the National Tonsil Surgery Register in Sweden. Clin Otolaryngol. 2015 Jun;40(3):248-54. doi: 10.1111/coa.12361. PMID 25515059
- [Background] Inuzuka Y, Mizutari K, Kamide D, Sato M, Shiotani A. Risk factors of post-tonsillectomy hemorrhage in adults. Laryngoscope Investig Otolaryngol. 2020 Nov 14;5(6):1056-1062. doi: 10.1002/lio2.488. eCollection 2020 Dec. PMID 33364394
- [Derived] Xu H, Qiu S, Pu S, Hu B, Liu D, Li X. Multicentre clinical study of haemorrhage after coblation tonsillectomy in children: a prospective study protocol. BMJ Open. 2023 Jan 10;13(1):e063401. doi: 10.1136/bmjopen-2022-063401. PMID 36627154